CLINICAL TRIAL: NCT03209908
Title: The Study of Starting to Use Tenofovir Disoproxil Fumarate(TDF) Antiviral Treatment From the 32 Weeks of Gestation to Block Mother-to-child Transmission of Hepatitis B Virus(HBV MTCT) and Withdrawal Time
Brief Title: The Study of Short-range Antiviral Treatment During Pregnancy to Block Mother-to-child Transmission of Hepatitis B Virus and Withdrawal Time
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Other Study IDs: XMLX201706-1
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis B
Keywords: antiviral treatment; hepatitis B virus; mother-to-child transmission; Tenofovir Disoproxil Fumarate
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the age of seven months, we extract venous blood of these children, separate the serums and collect the PBMC. Then, the serums are applied to test HBsAg, AntiHBs and HBVDNA which we adopt to analyse HLA classⅠand class Ⅱ gene polymorphism. meanwhile, detect HBVDNA loads of pregnant women with HBsAg/HBeAg positive and HBV DNA > 106 copies/ml in 32 weeks，36 weeks of gestation and before delivery.

GROUPS / COHORTS (2):
- control group: In this group, pregnant women with HBsAg/HBeAg positive and HBV DNA > 106 copies/ml don not use any antiviral drugs during pregnancy.
- experimental group: pregnant women with HBsAg/HBeAg positive and HBV DNA > 106 copies/ml start to use Tenofovir Disoproxil Fumarate(TDF) antiviral treatment from the 32 weeks of gestation to block mother-to-child transmission of hepatitis B virus.
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Tenofovir Disoproxil Fumarate was used for the experimental group of pregnancy women in the 32 weeks during pregnancy
  Other Names: TDF
  Groups: experimental group

SUMMARY:
Pregnant women carry high HBV DNA loads before delivery, which is the most important factor leading to mother-to-child transmission of HBV. Nucleoside analogue antiviral treatment during late pregnancy can significantly reduce the incidence of HBV MTCT, but security problems of using NA treatment during pregnancy has not been eliminated, Therefore, the aim of our study is to explore the effect of starting to use Tenofovir Disoproxil Fumarate(TDF) antiviral treatment from the 32 weeks of gestation to block mother-to-child transmission of hepatitis B virus(HBV MTCT).

DETAILED DESCRIPTION:
HBV MTCT is the important reason to keep high prevalence of chronic HBV infection in China; high HBV DNA loads of Pregnant women before delivery is the most important factor resulting in mother-to-child transmission of HBV, therefore, how to drop HBV DNA levels of pregnant women before delivery to the level that can markedly decrease the rate of HBV MTCT on the base of HBIG combined hepatitis b vaccine injection for newborns, which is the most important method to improve HBV MTCT. Although Nucleoside analogue antiviral treatment during late pregnancy can dramatically reduce the rate of HBV MTCT, security problems of NA treatment during pregnancy has not been demonstrated, On account of the above problems, our study is to investigate the effect of starting to use Tenofovir Disoproxil Fumarate(TDF) antiviral treatment from the 32 weeks of gestation to block mother-to-child transmission of hepatitis B virus(HBV MTCT).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were chronic hepatitis B and had achieved HBeAg positive and HBV DNA > 106 copies/ml

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus, HIV, etc.
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver
* without gestational hypertension, premature rupture of membranes, antepartum haemorrhage diseases or amniotic fluid piercing history during pregnancy.

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: In this study,the study population were composed of pregnant women suffering from chronic hepatitis B who had achieved HBsAg/HBeAg positive and HBV DNA > 106 copies/ml
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2017-01-01; Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
the blocking rate of vertical transmission of hepatitis B | seven months
  At the birth of 7 months, the venous blood serum HBsAg positive was defined as the failure of the interruption of HBV mother-to-child transmission.

SECONDARY OUTCOMES:
anti HBs level at the age of one month and seven months | one month and seven months
  Observing the level of anti HBs, then discussing the efficiency of personalized blocking method of HBV maternal-neonatal transmission

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China